CLINICAL TRIAL: NCT03103061
Title: Use of Lexiscan for Myocardial Stress Perfusion Computed Tomography With a 3rd Generation Dual Source CT System
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Collaborators: Astellas Pharma US, Inc. (Industry)
Responsible Party: Principal Investigator, U. Joseph Schoepf, MD, Professor, Medical University of South Carolina
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: Pro00051308
Record Dates: First submitted 2017-03-28; First posted 2017-04-06 (Actual); Results first posted 2019-08-09 (Actual); Last update posted 2019-08-09 (Actual); Status verified 2019-07

CONDITIONS: Cardiovascular Diseases; Coronary Artery Disease
Keywords: Computed Tomography
MeSH Terms: conditions — Cardiovascular Diseases; Coronary Artery Disease | interventions — regadenoson

STUDY DESIGN:
Intervention Model Description: Stress and rest perfusion imaging using Lexiscan as the coronary vasodilator (pharmacological stressor).

ARMS (1):
- Myocardial Stress CT Perfusion (Experimental): Low-radiation, dynamic perfusion CT of the heart in patients with suspected ischemic chest pain and a moderate or severe stenosis seen on coronary CTA. Lexiscan(TM) will be used as the pharmacological stress agent (coronary vasodilator).
  Interventions: Drug: Lexiscan

INTERVENTIONS:
Drug: Lexiscan — Coronary vasodilator

SUMMARY:
The purpose of this study is to evaluate the feasibility, tolerability, safety, and image quality of low-radiation, dynamic perfusion CT of the heart in patients with suspected ischemic chest pain and a moderate or severe stenosis seen on coronary CTA. Secondary aims include the assessment of the diagnostic accuracy of CT perfusion imaging compared to either SPECT or invasive angiography.

ELIGIBILITY:
Inclusion Criteria:

1. Subject must present with symptoms (e.g. chest pain) suspicious for cardiac ischemia as determined by treating physician.
2. Subject must have been referred for cardiac CT angiography OR subject must have undergone clinically indicated SPECT with positive or equivocal findings OR subject must have undergone clinically indicated SPECT with prior cardiac CT angiography that showed moderate or severe stenosis.
3. Subject must be 18 - 85 years of age.
4. Subject must provide written informed consent prior to any study-related procedures being performed.
5. Subject must be willing to comply with all clinical study procedures.

Exclusion Criteria:

1. Subject is a pregnant or nursing female. Exclude the possibility of pregnancy:

   * By testing (serum or urine beta HCG) within 24 hours before study agent administration, or
   * By surgical sterilization, or
   * Post menopausal, with minimum one (1) year history without menses.
2. Subject has severe asthma or COPD requiring frequent inhaler use.
3. Subject has prior diagnosis of obstructive CAD that has not been revascularized.
4. Subject with implanted rhythm devices (pacemaker, defibrillator).
5. Subject has significant arrhythmia.
6. Subject has high grade heart block.
7. Subject has resting heart rate < 45 bpm, systolic blood pressure <90 mm Hg, or has consumed caffeine within the last 12 hours.
8. Subject has an acute psychiatric disorder.
9. Subject is unwilling to comply with the requirements of the protocol.
10. Subject has previously entered this study.
11. Subject has an allergy against iodinated contrast agents or pharmaceutical stressors used in this study.
12. Subject suffers from claustrophobia.
13. Subject has impaired renal function (creatinine > 1.5 mg/dl).
14. Subject is in unstable condition.
15. ST-elevations, new transient ST changes greater than 0.05mV or T- wave inversions with symptoms
16. Subject cannot safely be administered Lexiscan™ per prescribing information as determined by investigator
17. Subject has received interventional (PCI, stenting) or surgical (CABG) treatment that may alter the cardiac condition regarding myocardial perfusion status and/or stenosis degree between cardiac CTA, SPECT, and/or CT stress perfusion studies.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2016-02-09 (Actual); Primary Completion 2018-06-14 (Actual); Study Completion 2018-06-14 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Medical University of South Carolina, Charleston, South Carolina, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Standard Subject Enrollment: Patients will undergo dynamic, stress perfusion computed tomography imaging during maximal hyperemia induced with Lexiscan™. CT MPI studies will use 40 - 50 mL of contrast agent (Ultravist 370) administered at a flow rate of 4 - 6 mL/s. Following the perfusion imaging, the Lexiscan™ will be reversed with 1 mg/kg of aminophylline per standard clinical protocol if indicated by the supervising physician.
Period: Overall Study
Arm/Group | Standard Subject Enrollment
Started | 24
Completed | 24
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Standard Subject Enrollment
Number analyzed (Participants) | 24
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 24
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17
  Male | 7
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 6
  White | 18
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 24

OUTCOME MEASURES:

1. Primary Outcome: Number of Treatment-related Adverse Events
Description: Demonstrate that CTA with stress and rest perfusion imaging using Lexiscan as the coronary vasodilator will be safe and well tolerated.
  This outcome measure data value represents the number of adverse events that occurred during this study.
Time Frame: 30 days +/- 3 days
Measure: Number; unit: Adverse events
Arm/Group | Standard Subject Enrollment
Number analyzed (Participants) | 24
Adverse events | 6

2. Secondary Outcome: Diagnostic Accuracy Using Quantitative Objective Image Quality Assessment
Description: Assess the diagnostic accuracy of CT perfusion imaging compared to either SPECT or invasive angiography.
Time Frame: Immediately following CT perfusion imaging.
Measure: Number; unit: Percent
Arm/Group | Standard Subject Enrollment
Number analyzed (Participants) | 24
Percent
  Sensitivity | 85.7
  Specificity | 70.6
  Accuracy | 75

ADVERSE EVENTS:
Time Frame: 30 days +/- 3 days
Groups:
- Standard Subject Enrollment: This study will plan to include 100 adults who present to the MUSC ED, hospital, or outpatient clinic with a clinical history and symptoms suspicious for cardiac ischemia and who have undergone or will likely undergo nuclear stress testing (SPECT).
  Patients who have been referred for a coronary CTA performed as part of a standard clinical evaluation determined by the treating physician(s) will be eligible for the study and recruited from the MUSC CT schedule. Before the patient comes in for their clinical coronary CTA, their cardiologist or primary physician will be contacted to ensure patient interest in the study and willingness to be approached. Willing patients will be approached and will undergo the informed consent process.
Arm/Group | Standard Subject Enrollment
All-Cause Mortality (participants affected / at risk) | 0/24
Serious Adverse Events (participants affected / at risk) | 0/24
Other Adverse Events (participants affected / at risk) | 0/24

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-05-11): https://cdn.clinicaltrials.gov/large-docs/61/NCT03103061/Prot_SAP_000.pdf